CLINICAL TRIAL: NCT02568215
Title: A Phase 2b Study to Evaluate the Safety and Efficacy of VRC01 Broadly Neutralizing Monoclonal Antibody in Reducing Acquisition of HIV-1 Infection in Women in Sub-Saharan Africa
Brief Title: Evaluating the Safety and Efficacy of the VRC01 Antibody in Reducing Acquisition of HIV-1 Infection in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 703/HPTN 081; 12045 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: HIV Infections
Keywords: HIV-1 Infections
MeSH Terms: conditions — HIV Infections | interventions — VRC01 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: Low-Dose VRC01 (Experimental): Participants will receive an IV infusion of 10 mg/kg of VRC01 over about 30 to 60 minutes at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, and 72.
  Interventions: Biological: VRC01
- Group 2: High-Dose VRC01 (Experimental): Participants will receive an IV infusion of 30 mg/kg of VRC01 over about 30 to 60 minutes at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, and 72.
  Interventions: Biological: VRC01
- Group 3: Placebo for VRC01 (Placebo Comparator): Participants will receive an IV infusion of placebo for VRC01 over about 30 to 60 minutes at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, and 72.
  Interventions: Biological: Placebo for VRC01

INTERVENTIONS:
Biological: VRC01 — Administered by IV infusion; total dose will vary based on participant's weight
  Other Names: Human monoclonal antibody (mAb) VRC-HIVMAB060-00-AB
  Arms: Group 1: Low-Dose VRC01; Group 2: High-Dose VRC01
Biological: Placebo for VRC01 — Sodium Chloride for Injection USP, 0.9%; administered by IV infusion
  Arms: Group 3: Placebo for VRC01

SUMMARY:
This study will evaluate the safety and efficacy of the human monoclonal antibody (mAb) VRC-HIVMAB060-00-AB (VRC01) in preventing HIV-1 infection in high-risk, HIV-uninfected women.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and efficacy of the VRC01 antibody in preventing HIV-1 infection in healthy women at high risk of HIV infection.

Participants will be enrolled from a cohort of heterosexual women in sub-Saharan Africa. An equal number of study participants will be randomized to receive VRC01 mAb by IV infusion at a dose of 10 mg/kg or 30 mg/kg every 8 weeks, or to receive control infusions every 8 weeks. All participants will receive the VRC01 antibody or placebo by intravenous infusion at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72. For 3 days following each infusion, participants will be asked to record and report any symptoms to study researchers.

In addition to the infusion visits, participants will attend study visits at Weeks 4, 8 + 5 days, 12, 20, 28, 36, 44, 52, 60, 68, 76, 80, 84, 88, and 92. All study visits will include blood collection and HIV testing and counseling. Select study visits will include a medical history review, physical exam, urine collection, pregnancy testing for participants capable of becoming pregnant, risk reduction counseling, and an interview/questionnaire.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study and completes a questionnaire prior to first infusion with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent for the duration of the participant's trial participation
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Persons born Female (assigned female sex at birth) and identifying as a female, who, in the 6 months prior to randomization, has had vaginal and/or anal intercourse with a male partner
* All volunteers who have been in a monogamous relationship with an HIV-1 seronegative partner for greater than 1 year are excluded.

Laboratory Inclusion Values+

Hematology

* Hemoglobin (Hgb) greater than or equal to 10.5 g/dL for volunteers who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male
* Platelets greater than or equal to 100,000 cells/mm^3

Chemistry

* Alanine aminotransferase (ALT) less than 2.5 times the institutional upper limit of normal and creatinine less than or equal to 1.25 times the institutional upper limit of normal

Virology

* HIV uninfected, as defined in the study specific procedures (SSP), within 30 days prior to enrollment

Urine

* Negative, trace, or 1+ urine protein by dipstick

Reproductive Status

* Volunteers capable of becoming pregnant: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed at the screening visit and prior to infusion on the day of initial infusion. Persons who are NOT capable of becoming pregnant due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records) are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who is capable of becoming pregnant must agree to consistently use effective contraception (see the protocol and SSP for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit.
* Volunteers capable of becoming pregnant must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General

* Investigational research agents received within 30 days before first infusion
* Body mass index (BMI) greater than or equal to 40
* Pregnant or breastfeeding
* Any reactive, indeterminate, or positive HIV test, even if subsequent testing indicates that the individual is not HIV infected.

Monoclonal antibodies and vaccines

* Previous receipt of humanized or human monoclonal antibodies (mAbs), whether licensed or investigational
* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 703/HPTN 081 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.

Immune System

* Serious adverse reactions to VRC01 formulation components such as sodium citrate, sodium chloride, and L-arginine hydrochloride, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain.
* Autoimmune disease, including Type I diabetes mellitus (Not excluded from participation: Volunteer with mild, stable and uncomplicated autoimmune disease that does not require consistent immunosuppressive medication and that, in the judgment of the site investigator, is likely not subject to exacerbation and likely not to complicate reactogenicity and adverse event (AE) assessments)
* Immunodeficiency syndrome

Clinically significant medical conditions

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * Any contraindication to repeated infusions or blood draws, including inability to establish venous access;
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period; or
  * A condition or process for which signs or symptoms could be confused with reactions to VRC01.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or infusion reactions, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Asthma, other than mild, well-controlled asthma
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure. or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema
* History of organ or tissue transplantation
* Known hepatic or renal dysfunction

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1924 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Corey, Study Chair — HVTN; FHCRC; Myron Cohen, Study Chair — HPTN; University of North Carolina
Locations (21):
- Gaborone CRS, Gaborone, South-East District, Botswana
- Kisumu Crs, Kisumu, Nyanza, Kenya
- Malawi (2):
  - Blantyre CRS, Blantyre, Southern Region
  - Malawi CRS, Lilongwe
- Polana Canico Health Research and Training Center (CISPOC), National Institute of Health (INS) CRS, Maputo, Mozambique
- South Africa (12):
  - The Aurum Institute Tembisa Clinical Research Centre CRS, Johannesburg, Gauteng
  - Soweto HVTN CRS, Johannesburg, Gauteng
  - Ward 21 CRS, Johannesburg, Gauteng
  - Wits Reproductive Health and HIV Institute CRS (WRHI CRS), Johannesburg, Gauteng
  - Synexus Stanza Clinical Research Centre CRS, Pretoria, Gauteng
  - Chatsworth CRS, Chatsworth, KwaZulu-Natal
  - Botha's Hill CRS, Durban, KwaZulu-Natal
  - CAPRISA eThekwini CRS, Durban, KwaZulu-Natal
  - Vulindlela CRS, Durban, KwaZulu-Natal
  - Aurum Institute Klerksdorp CRS, Klerksdorp, North West
  - Rustenburg CRS, Rustenburg, North West
  - Groote Schuur HIV CRS, Cape Town, Western Cape
- National Institute for Medical Research (NIMR) - Mbeya Medical Research Center (MMRC) Network CRS, Mbeya, Tanzania
- Zimbabwe (3):
  - Seke South CRS, Chitungwiza
  - Milton Park CRS, Harare
  - Spilhaus CRS, Harare

REFERENCES:
- [Result] Edupuganti S, Mgodi N, Karuna ST, Andrew P, Rudnicki E, Kochar N, deCamp A, De La Grecca R, Anderson M, Karg C, Tindale I, Greene E, Broder GB, Lucas J, Hural J, Gallardo-Cartagena JA, Gonzales P, Frank I, Sobieszczyk M, Gomez Lorenzo MM, Burns D, Anderson PL, Miner MD, Ledgerwood J, Mascola JR, Gilbert PB, Cohen MS, Corey L; HVTN 704/HPTN 085 study group. Feasibility and Successful Enrollment in a Proof-of-Concept HIV Prevention Trial of VRC01, a Broadly Neutralizing HIV-1 Monoclonal Antibody. J Acquir Immune Defic Syndr. 2021 May 1;87(1):671-679. doi: 10.1097/QAI.0000000000002639. PMID 33587505
- [Result] Mgodi NM, Takuva S, Edupuganti S, Karuna S, Andrew P, Lazarus E, Garnett P, Shava E, Mukwekwerere PG, Kochar N, Marshall K, Rudnicki E, Juraska M, Anderson M, Karg C, Tindale I, Greene E, Luthuli N, Baepanye K, Hural J, Gomez Lorenzo MM, Burns D, Miner MD, Ledgerwood J, Mascola JR, Donnell D, Cohen MS, Corey L; HVTN 703/HPTN 081 Team. A Phase 2b Study to Evaluate the Safety and Efficacy of VRC01 Broadly Neutralizing Monoclonal Antibody in Reducing Acquisition of HIV-1 Infection in Women in Sub-Saharan Africa: Baseline Findings. J Acquir Immune Defic Syndr. 2021 May 1;87(1):680-687. doi: 10.1097/QAI.0000000000002649. PMID 33587510
- [Result] Huang Y, Naidoo L, Zhang L, Carpp LN, Rudnicki E, Randhawa A, Gonzales P, McDermott A, Ledgerwood J, Lorenzo MMG, Burns D, DeCamp A, Juraska M, Mascola J, Edupuganti S, Mgodi N, Cohen M, Corey L, Andrew P, Karuna S, Gilbert PB, Mngadi K, Lazarus E. Pharmacokinetics and predicted neutralisation coverage of VRC01 in HIV-uninfected participants of the Antibody Mediated Prevention (AMP) trials. EBioMedicine. 2021 Feb;64:103203. doi: 10.1016/j.ebiom.2020.103203. Epub 2021 Jan 23. PMID 33493795
- [Result] Huang Y, Zhang L, Eaton A, Mkhize NN, Carpp LN, Rudnicki E, DeCamp A, Juraska M, Randhawa A, McDermott A, Ledgerwood J, Andrew P, Karuna S, Edupuganti S, Mgodi N, Cohen M, Corey L, Mascola J, Gilbert PB, Morris L, Montefiori DC. Prediction of serum HIV-1 neutralization titers of VRC01 in HIV-uninfected Antibody Mediated Prevention (AMP) trial participants. Hum Vaccin Immunother. 2022 Dec 31;18(1):1908030. doi: 10.1080/21645515.2021.1908030. Epub 2021 Jul 2. PMID 34213402
- [Result] Corey L, Gilbert PB, Juraska M, Montefiori DC, Morris L, Karuna ST, Edupuganti S, Mgodi NM, deCamp AC, Rudnicki E, Huang Y, Gonzales P, Cabello R, Orrell C, Lama JR, Laher F, Lazarus EM, Sanchez J, Frank I, Hinojosa J, Sobieszczyk ME, Marshall KE, Mukwekwerere PG, Makhema J, Baden LR, Mullins JI, Williamson C, Hural J, McElrath MJ, Bentley C, Takuva S, Gomez Lorenzo MM, Burns DN, Espy N, Randhawa AK, Kochar N, Piwowar-Manning E, Donnell DJ, Sista N, Andrew P, Kublin JG, Gray G, Ledgerwood JE, Mascola JR, Cohen MS; HVTN 704/HPTN 085 and HVTN 703/HPTN 081 Study Teams. Two Randomized Trials of Neutralizing Antibodies to Prevent HIV-1 Acquisition. N Engl J Med. 2021 Mar 18;384(11):1003-1014. doi: 10.1056/NEJMoa2031738. PMID 33730454
- [Derived] Reeves DB, Mayer BT, deCamp AC, Huang Y, Zhang B, Carpp LN, Magaret CA, Juraska M, Gilbert PB, Montefiori DC, Bar KJ, Cardozo-Ojeda EF, Schiffer JT, Rossenkhan R, Edlefsen P, Morris L, Mkhize NN, Williamson C, Mullins JI, Seaton KE, Tomaras GD, Andrew P, Mgodi N, Ledgerwood JE, Cohen MS, Corey L, Naidoo L, Orrell C, Goepfert PA, Casapia M, Sobieszczyk ME, Karuna ST, Edupuganti S. High monoclonal neutralization titers reduced breakthrough HIV-1 viral loads in the Antibody Mediated Prevention trials. Nat Commun. 2023 Dec 14;14(1):8299. doi: 10.1038/s41467-023-43384-y. PMID 38097552
- [Derived] Hanass-Hancock J, Carpenter B, Reddy T, Nzuza A, Gaffoor Z, Goga A, Andrasik M. Participants' characteristics and motivations to screen for HIV vaccine and monoclonal antibody trials in KwaZulu-Natal, South Africa. Trials. 2021 Dec 11;22(1):897. doi: 10.1186/s13063-021-05792-7. PMID 34895272

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned to the placebo, low-dose VRC01, or high-dose VRC01 arm. The pooled VRC01 arm represents participants assigned to low-dose or high-dose VRC01 and is the primary comparison group for the primary analysis of prevention efficacy.
Groups:
- Placebo: Placebo (Sodium Chloride, USP 0.9%) by intravenous (IV) infusion at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72.
- Low-Dose VRC01: VRC01 mAb by intravenous (IV) infusion at a dose of 10 mg/kg at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72.
- High-Dose VRC01: VRC01 mAb by intravenous (IV) infusion at a dose of 30 mg/kg at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72.
Period: Overall Study
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01
Started (Enrollment is concurrent with receiving the first infusion (safety analyses)) | 637 | 642 | 645
Modified Intent-to-treat Population (Participants excluded from MITT if HIV positive at enrollment or randomized/enrolled more than once (efficacy analyses)) | 637 | 642 | 645
Completed | 558 | 562 | 555
Not Completed | 79 | 80 | 90
Not completed — Death | 1 | 2 | 0
Not completed — Physician Decision | 2 | 2 | 2
Not completed — Lost to Follow-up | 29 | 32 | 41
Not completed — Withdrawal by Subject | 21 | 19 | 22
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Participant Unable to Adhere to Visit Schedule | 25 | 23 | 21
Not completed — Other | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Total
Number analyzed (Participants) | 637 | 642 | 645 | 1924
Age, Continuous [Median (Full Range); unit: years] | 26 [18 to 45] | 25 [17 to 43] | 26 [18 to 44] | 25 [17 to 45]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 1 | 0 | 1
  18 - 20 years | 84 | 86 | 89 | 259
  21 - 30 years | 408 | 416 | 411 | 1235
  31 - 40 years | 142 | 136 | 142 | 420
  41 - 50 years | 3 | 3 | 3 | 9
  Above 50 years | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 637 | 642 | 645 | 1924
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 637 | 642 | 645 | 1924
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 0 | 0 | 0
  Black | 628 | 635 | 639 | 1902
  Asian | 0 | 0 | 0 | 0
  Indian | 5 | 1 | 3 | 9
  Colored/Mixed | 3 | 6 | 3 | 12
  More than one race | 1 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Mozambique | 8 | 9 | 9 | 26
  Malawi | 59 | 60 | 61 | 180
  Botswana | 47 | 52 | 51 | 150
  Tanzania | 11 | 12 | 10 | 33
  South Africa | 340 | 338 | 341 | 1019
  Zimbabwe | 145 | 144 | 145 | 434
  Kenya | 27 | 27 | 28 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented
Time Frame: Measured through 3 days after each infusion at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Pooled VRC01: VRC01 mAb by intravenous (IV) infusion at a dose of 10 or 30 mg/kg at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72.
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
Participants
  Pain: None | 476 | 496 | 506 | 1002
  Pain: Mild | 142 | 120 | 120 | 240
  Pain: Moderate | 19 | 26 | 16 | 42
  Pain: Severe | 0 | 0 | 3 | 3
  Pain: Potentially Life-threatening | 0 | 0 | 0 | 0
  Tenderness: None | 518 | 547 | 543 | 1090
  Tenderness: Mild | 104 | 81 | 87 | 168
  Tenderness: Moderate | 15 | 13 | 13 | 26
  Tenderness: Severe | 0 | 1 | 2 | 3
  Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 452 | 482 | 476 | 958
  Pain and/or Tenderness: Mild | 162 | 133 | 144 | 277
  Pain and/or Tenderness: Moderate | 23 | 26 | 22 | 48
  Pain and/or Tenderness: Severe | 0 | 1 | 3 | 4
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through 3 days after each infusion at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
Participants
  Erythema/Redness: None or Not Gradable | 618 | 618 | 629 | 1247
  Erythema/Redness: Gr 1: 6.25 to less than 25 sq.cm or 2.5 to less than 5 cm single dim. | 12 | 17 | 12 | 29
  Erythema/Redness: Gr 2: 25 to less than 100 sq.cm or 5 to less than 10 cm single dim. | 7 | 7 | 4 | 11
  Erythema/Redness: Gr 3: >=100 sq.cm or >=10 cm single dim or severe complication | 0 | 0 | 0 | 0
  Erythema/Redness: Gr 4: Potentially Life-Threatening complication | 0 | 0 | 0 | 0
  Induration/Swelling: None or Not Gradable | 623 | 632 | 639 | 1271
  Induration/Swelling: Gr 1: 6.25 to less than 25 sq.cm or 2.5 to less than 5 cm single dim. | 12 | 9 | 5 | 14
  Induration/Swelling: Gr 2: 25 to less than 100 sq.cm or 5 to less than 10 cm single dim. | 2 | 1 | 1 | 2
  Induration/Swelling: Gr 3: >=100 sq.cm or >=10 cm single dim or severe complication | 0 | 0 | 0 | 0
  Induration/Swelling: Gr 4: Potentially Life-Threatening complication | 0 | 0 | 0 | 0
  Erythema and/or Induration: None or Not Gradable | 610 | 612 | 627 | 1239
  Erythema and/or Induration: Gr 1: 6.25 to less than 25 sq.cm or 2.5 to less than 5 cm single dim. | 20 | 22 | 13 | 35
  Erythema and/or Induration: Gr 2: 25 to less than 100 sq.cm or 5 to less than 10 cm single dim. | 7 | 8 | 5 | 13
  Erythema and/or Induration: Gr 3: >=100 sq.cm or >=10 cm single dim or severe complication | 0 | 0 | 0 | 0
  Erythema and/or Induration: Gr 4: Potentially Life-Threatening complication | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The following symptoms are considered as systemic reactogenicity if the onset date was within the periods of assessment specified in the protocol: malaise and/or fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and body temperature. The item Max. Systemic Symptoms is the maximum of the individual systemic reactogenicities excluding body temperature for a participant.
Time Frame: Measured through 3 days after each infusion at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
Participants
  Malaise and/or fatigue: None | 473 | 487 | 495 | 982
  Malaise and/or fatigue: Mild | 134 | 122 | 107 | 229
  Malaise and/or fatigue: Moderate | 30 | 33 | 42 | 75
  Malaise and/or fatigue: Severe | 0 | 0 | 1 | 1
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0
  Myalgia: None | 561 | 574 | 579 | 1153
  Myalgia: Mild | 57 | 50 | 54 | 104
  Myalgia: Moderate | 19 | 18 | 12 | 30
  Myalgia: Severe | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Headache: None | 382 | 394 | 387 | 781
  Headache: Mild | 198 | 182 | 188 | 370
  Headache: Moderate | 57 | 66 | 70 | 136
  Headache: Severe | 0 | 0 | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0
  Nausea: None | 549 | 565 | 567 | 1132
  Nausea: Mild | 76 | 70 | 65 | 135
  Nausea: Moderate | 12 | 7 | 13 | 20
  Nausea: Severe | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0
  Vomiting: None | 603 | 611 | 614 | 1225
  Vomiting: Mild | 26 | 28 | 28 | 56
  Vomiting: Moderate | 8 | 3 | 3 | 6
  Vomiting: Severe | 0 | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0
  Chills: None | 589 | 591 | 599 | 1190
  Chills: Mild | 40 | 43 | 37 | 80
  Chills: Moderate | 8 | 8 | 9 | 17
  Chills: Severe | 0 | 0 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0
  Arthralgia: None | 577 | 576 | 596 | 1172
  Arthralgia: Mild | 43 | 54 | 36 | 90
  Arthralgia: Moderate | 17 | 12 | 13 | 25
  Arthralgia: Severe | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 319 | 328 | 326 | 654
  Max. Systemic Symptoms: Mild | 246 | 230 | 233 | 463
  Max. Systemic Symptoms: Moderate | 72 | 84 | 85 | 169
  Max. Systemic Symptoms: Severe | 0 | 0 | 1 | 1
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0
  Increased Body Temperature: None | 609 | 610 | 616 | 1226
  Increased Body Temperature: Mild | 15 | 14 | 20 | 34
  Increased Body Temperature: Moderate | 10 | 16 | 7 | 23
  Increased Body Temperature: Severe | 3 | 2 | 2 | 4
  Increased Body Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0

4. Primary Outcome: Chemistry and Hematology Laboratory Measures - Alanine Aminotransferase (ALT)
Description: For each local laboratory measure, summary statistics are presented by treatment group and timepoint.
Time Frame: Measured at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: Safety population. Participants may not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
U/L
  ALT (SGPT) (U/L)- Week 0: number analyzed (Participants) | 636 | 642 | 645 | 1287
  ALT (SGPT) (U/L)- Week 0 | 15 [12 to 21] | 15 [12 to 20] | 16 [12 to 22] | 15 [12 to 21]
  ALT (SGPT) (U/L)- Week 8: number analyzed (Participants) | 618 | 612 | 608 | 1220
  ALT (SGPT) (U/L)- Week 8 | 15 [12 to 21] | 15 [11 to 20] | 16 [12 to 22] | 15 [12 to 21]
  ALT (SGPT) (U/L)- Week 16: number analyzed (Participants) | 606 | 593 | 589 | 1182
  ALT (SGPT) (U/L)- Week 16 | 16 [12 to 22] | 15 [11 to 20] | 16 [12 to 21] | 15 [12 to 21]
  ALT (SGPT) (U/L)- Week 24: number analyzed (Participants) | 594 | 587 | 581 | 1168
  ALT (SGPT) (U/L)- Week 24 | 16 [12 to 22] | 14 [11 to 20] | 16 [12 to 21] | 15 [12 to 21]
  ALT (SGPT) (U/L)- Week 32: number analyzed (Participants) | 577 | 568 | 572 | 1140
  ALT (SGPT) (U/L)- Week 32 | 16 [12 to 22] | 15 [12 to 21] | 16 [12 to 21.5] | 16 [12 to 21]
  ALT (SGPT) (U/L)- Week 40: number analyzed (Participants) | 563 | 554 | 554 | 1108
  ALT (SGPT) (U/L)- Week 40 | 16 [12 to 23] | 15 [11 to 21] | 15 [12 to 22] | 15 [12 to 21]
  ALT (SGPT) (U/L)- Week 48: number analyzed (Participants) | 560 | 542 | 539 | 1081
  ALT (SGPT) (U/L)- Week 48 | 16 [12 to 22] | 15 [12 to 21] | 16 [12 to 21] | 15 [12 to 21]
  ALT (SGPT) (U/L)- Week 56: number analyzed (Participants) | 553 | 533 | 538 | 1071
  ALT (SGPT) (U/L)- Week 56 | 16 [12 to 22] | 15 [12 to 20] | 16 [12 to 21] | 16 [12 to 21]
  ALT (SGPT) (U/L)- Week 64: number analyzed (Participants) | 548 | 530 | 536 | 1066
  ALT (SGPT) (U/L)- Week 64 | 16 [12 to 22] | 15 [12 to 20] | 15 [12 to 21] | 15 [12 to 20]
  ALT (SGPT) (U/L)- Week 72: number analyzed (Participants) | 541 | 514 | 526 | 1040
  ALT (SGPT) (U/L)- Week 72 | 16 [12 to 21] | 15 [12 to 20] | 15 [12 to 20] | 15 [12 to 20]

5. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine
Description: For each local laboratory measure, summary statistics are presented by treatment group and timepoint.
Time Frame: Measured at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
mg/dL
  Creatinine (mg/dL)- Week 0: number analyzed (Participants) | 636 | 642 | 645 | 1287
  Creatinine (mg/dL)- Week 0 | 0.64 [0.59 to 0.72] | 0.66 [0.6 to 0.73] | 0.67 [0.59 to 0.72] | 0.66 [0.6 to 0.73]
  Creatinine (mg/dL)- Week 8: number analyzed (Participants) | 618 | 612 | 608 | 1220
  Creatinine (mg/dL)- Week 8 | 0.65 [0.59 to 0.73] | 0.66 [0.6 to 0.72] | 0.66 [0.59 to 0.73] | 0.66 [0.59 to 0.73]
  Creatinine (mg/dL)- Week 16: number analyzed (Participants) | 606 | 593 | 589 | 1182
  Creatinine (mg/dL)- Week 16 | 0.66 [0.6 to 0.72] | 0.66 [0.6 to 0.74] | 0.67 [0.6 to 0.75] | 0.67 [0.6 to 0.74]
  Creatinine (mg/dL)- Week 24: number analyzed (Participants) | 594 | 587 | 581 | 1168
  Creatinine (mg/dL)- Week 24 | 0.67 [0.6 to 0.74] | 0.68 [0.61 to 0.74] | 0.67 [0.6 to 0.74] | 0.67 [0.6 to 0.74]
  Creatinine (mg/dL)- Week 32: number analyzed (Participants) | 577 | 568 | 572 | 1140
  Creatinine (mg/dL)- Week 32 | 0.66 [0.6 to 0.74] | 0.67 [0.6 to 0.74] | 0.67 [0.6 to 0.75] | 0.67 [0.6 to 0.75]
  Creatinine (mg/dL)- Week 40: number analyzed (Participants) | 563 | 554 | 554 | 1108
  Creatinine (mg/dL)- Week 40 | 0.67 [0.6 to 0.75] | 0.67 [0.6 to 0.75] | 0.68 [0.6 to 0.75] | 0.67 [0.6 to 0.75]
  Creatinine (mg/dL)- Week 48: number analyzed (Participants) | 560 | 542 | 539 | 1081
  Creatinine (mg/dL)- Week 48 | 0.67 [0.59 to 0.75] | 0.67 [0.6 to 0.75] | 0.68 [0.61 to 0.75] | 0.68 [0.6 to 0.75]
  Creatinine (mg/dL)- Week 56: number analyzed (Participants) | 553 | 533 | 538 | 1071
  Creatinine (mg/dL)- Week 56 | 0.67 [0.6 to 0.74] | 0.67 [0.61 to 0.76] | 0.68 [0.61 to 0.75] | 0.68 [0.61 to 0.76]
  Creatinine (mg/dL)- Week 64: number analyzed (Participants) | 548 | 530 | 536 | 1066
  Creatinine (mg/dL)- Week 64 | 0.67 [0.61 to 0.75] | 0.68 [0.6 to 0.75] | 0.68 [0.62 to 0.76] | 0.68 [0.61 to 0.75]
  Creatinine (mg/dL)- Week 72: number analyzed (Participants) | 541 | 514 | 526 | 1040
  Creatinine (mg/dL)- Week 72 | 0.67 [0.61 to 0.74] | 0.68 [0.61 to 0.74] | 0.68 [0.61 to 0.75] | 0.68 [0.61 to 0.75]

6. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin
Description: For each local laboratory measure, summary statistics are presented by treatment group and timepoint.
Time Frame: Measured at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
g/dL
  Hemoglobin (g/dL)- Week 0: number analyzed (Participants) | 637 | 642 | 642 | 1284
  Hemoglobin (g/dL)- Week 0 | 13.4 [12.6 to 14.2] | 13.4 [12.7 to 14.2] | 13.6 [12.8 to 14.3] | 13.5 [12.7 to 14.3]
  Hemoglobin (g/dL)- Week 8: number analyzed (Participants) | 618 | 610 | 608 | 1218
  Hemoglobin (g/dL)- Week 8 | 13.2 [12.6 to 13.9] | 13.2 [12.5 to 13.9] | 13.3 [12.45 to 14.1] | 13.2 [12.5 to 14]
  Hemoglobin (g/dL)- Week 16: number analyzed (Participants) | 606 | 593 | 586 | 1179
  Hemoglobin (g/dL)- Week 16 | 13.2 [12.4 to 13.9] | 13.1 [12.2 to 13.9] | 13.2 [12.3 to 13.9] | 13.1 [12.3 to 13.9]
  Hemoglobin (g/dL)- Week 24: number analyzed (Participants) | 594 | 586 | 581 | 1167
  Hemoglobin (g/dL)- Week 24 | 13.1 [12.4 to 13.9] | 13.1 [12.3 to 13.8] | 13.1 [12.4 to 13.9] | 13.1 [12.3 to 13.9]
  Hemoglobin (g/dL)- Week 32: number analyzed (Participants) | 576 | 567 | 574 | 1141
  Hemoglobin (g/dL)- Week 32 | 13.1 [12.3 to 13.9] | 13.1 [12.3 to 13.8] | 13.2 [12.3 to 13.9] | 13.1 [12.3 to 13.9]
  Hemoglobin (g/dL)- Week 40: number analyzed (Participants) | 564 | 554 | 556 | 1110
  Hemoglobin (g/dL)- Week 40 | 13.1 [12.3 to 13.9] | 13.15 [12.3 to 13.9] | 13.2 [12.3 to 14] | 13.2 [12.3 to 13.9]
  Hemoglobin (g/dL)- Week 48: number analyzed (Participants) | 559 | 543 | 539 | 1082
  Hemoglobin (g/dL)- Week 48 | 13 [12.3 to 13.9] | 13.1 [12.2 to 13.8] | 13.2 [12.4 to 13.9] | 13.1 [12.3 to 13.9]
  Hemoglobin (g/dL)- Week 56: number analyzed (Participants) | 553 | 533 | 538 | 1071
  Hemoglobin (g/dL)- Week 56 | 13.1 [12.3 to 13.9] | 13 [12.2 to 13.8] | 13.1 [12.4 to 13.8] | 13.1 [12.3 to 13.8]
  Hemoglobin (g/dL)- Week 64: number analyzed (Participants) | 545 | 529 | 537 | 1066
  Hemoglobin (g/dL)- Week 64 | 13 [12.3 to 13.8] | 13 [12.3 to 13.8] | 13.1 [12.4 to 13.9] | 13.1 [12.3 to 13.8]
  Hemoglobin (g/dL)- Week 72: number analyzed (Participants) | 540 | 515 | 526 | 1041
  Hemoglobin (g/dL)- Week 72 | 13 [12.15 to 13.8] | 13 [12.2 to 13.8] | 13.1 [12.3 to 13.9] | 13 [12.2 to 13.8]

7. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocyte Count, Neutrophil Count
Description: For each local laboratory measure, summary statistics are presented by treatment group and timepoint.
Time Frame: Measured at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: cells/cubic mm
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
cells/cubic mm
  Lymphocytes (cells/cubic mm)- Week 0: number analyzed (Participants) | 637 | 642 | 642 | 1284
  Lymphocytes (cells/cubic mm)- Week 0 | 2172 [1820 to 2560] | 2123 [1799 to 2540] | 2180 [1848 to 2570] | 2160 [1822 to 2560]
  Lymphocytes (cells/cubic mm)- Week 8: number analyzed (Participants) | 618 | 610 | 608 | 1218
  Lymphocytes (cells/cubic mm)- Week 8 | 2148 [1810 to 2490] | 2050 [1742 to 2424] | 2145.5 [1819.5 to 2514] | 2100 [1770 to 2478]
  Lymphocytes (cells/cubic mm)- Week 16: number analyzed (Participants) | 606 | 593 | 586 | 1179
  Lymphocytes (cells/cubic mm)- Week 16 | 2120 [1760 to 2487] | 2060 [1772 to 2408] | 2082.5 [1750 to 2450] | 2070 [1765 to 2430]
  Lymphocytes (cells/cubic mm)- Week 24: number analyzed (Participants) | 594 | 586 | 581 | 1167
  Lymphocytes (cells/cubic mm)- Week 24 | 2124.5 [1788 to 2460] | 2042 [1730 to 2400] | 2091 [1747 to 2472] | 2067 [1739 to 2428]
  Lymphocytes (cells/cubic mm)- Week 32: number analyzed (Participants) | 576 | 567 | 574 | 1141
  Lymphocytes (cells/cubic mm)- Week 32 | 2125.5 [1785 to 2489] | 2040 [1740 to 2449] | 2074.5 [1792 to 2470] | 2060 [1752 to 2458]
  Lymphocytes (cells/cubic mm)- Week 40: number analyzed (Participants) | 564 | 554 | 556 | 1110
  Lymphocytes (cells/cubic mm)- Week 40 | 2110.5 [1761.5 to 2457] | 2052 [1720 to 2451] | 2110 [1736 to 2470] | 2080 [1723 to 2459]
  Lymphocytes (cells/cubic mm)- Week 48: number analyzed (Participants) | 559 | 543 | 539 | 1082
  Lymphocytes (cells/cubic mm)- Week 48 | 2111 [1781 to 2448] | 2042 [1720 to 2396] | 2148 [1790 to 2504] | 2080 [1751 to 2457]
  Lymphocytes (cells/cubic mm)- Week 56: number analyzed (Participants) | 552 | 533 | 538 | 1071
  Lymphocytes (cells/cubic mm)- Week 56 | 2082.5 [1765 to 2460.5] | 2000 [1734 to 2400] | 2120.5 [1760 to 2487] | 2051 [1750 to 2436]
  Lymphocytes (cells/cubic mm)- Week 64: number analyzed (Participants) | 544 | 529 | 537 | 1066
  Lymphocytes (cells/cubic mm)- Week 64 | 2070 [1740 to 2434] | 2029 [1710 to 2379] | 2106 [1780 to 2470] | 2068.5 [1740 to 2430]
  Lymphocytes (cells/cubic mm)- Week 72: number analyzed (Participants) | 540 | 515 | 526 | 1041
  Lymphocytes (cells/cubic mm)- Week 72 | 2109.5 [1757 to 2459.5] | 2040 [1720 to 2420] | 2150 [1772 to 2447] | 2090 [1747 to 2431]
  Neutrophils (cells/cubic mm)- Week 0: number analyzed (Participants) | 637 | 642 | 642 | 1284
  Neutrophils (cells/cubic mm)- Week 0 | 3008 [2300 to 4113] | 2999 [2358 to 3950] | 3200 [2458 to 4147] | 3107.5 [2404.5 to 4051.5]
  Neutrophils (cells/cubic mm)- Week 8: number analyzed (Participants) | 618 | 610 | 608 | 1218
  Neutrophils (cells/cubic mm)- Week 8 | 2940.5 [2215 to 3930] | 2905.5 [2190 to 3750] | 3070 [2340 to 3980] | 2985 [2270 to 3859]
  Neutrophils (cells/cubic mm)- Week 16: number analyzed (Participants) | 606 | 593 | 586 | 1179
  Neutrophils (cells/cubic mm)- Week 16 | 2868.5 [2110 to 3834] | 2821 [2190 to 3760] | 3046.5 [2310 to 3976] | 2950 [2260 to 3900]
  Neutrophils (cells/cubic mm)- Week 24: number analyzed (Participants) | 594 | 586 | 581 | 1167
  Neutrophils (cells/cubic mm)- Week 24 | 2858 [2188 to 3930] | 2924 [2213 to 3800] | 2922 [2265 to 3960] | 2923 [2240 to 3900]
  Neutrophils (cells/cubic mm)- Week 32: number analyzed (Participants) | 576 | 567 | 574 | 1141
  Neutrophils (cells/cubic mm)- Week 32 | 2830 [2117.5 to 3863.5] | 2881 [2200 to 3969] | 2988 [2320 to 3931] | 2943 [2239 to 3956]
  Neutrophils (cells/cubic mm)- Week 40: number analyzed (Participants) | 564 | 554 | 556 | 1110
  Neutrophils (cells/cubic mm)- Week 40 | 2910 [2215 to 3939] | 2888.5 [2224 to 3779] | 3065 [2319 to 4062.5] | 3020.5 [2253 to 3905]
  Neutrophils (cells/cubic mm)- Week 48: number analyzed (Participants) | 559 | 543 | 539 | 1082
  Neutrophils (cells/cubic mm)- Week 48 | 2920 [2187 to 3910] | 2990 [2271 to 3908] | 2994 [2249 to 3956] | 2992.5 [2263 to 3930]
  Neutrophils (cells/cubic mm)- Week 56: number analyzed (Participants) | 552 | 533 | 538 | 1071
  Neutrophils (cells/cubic mm)- Week 56 | 3000 [2261 to 4045] | 2940 [2206 to 3846] | 2955.5 [2280 to 3830] | 2945 [2240 to 3846]
  Neutrophils (cells/cubic mm)- Week 64: number analyzed (Participants) | 544 | 529 | 537 | 1066
  Neutrophils (cells/cubic mm)- Week 64 | 2834 [2125 to 3908] | 2918 [2198 to 3862] | 2970 [2316 to 3870] | 2944 [2244 to 3866]
  Neutrophils (cells/cubic mm)- Week 72: number analyzed (Participants) | 540 | 515 | 526 | 1041
  Neutrophils (cells/cubic mm)- Week 72 | 2868.5 [2164.5 to 3836] | 2880 [2230 to 3726] | 2970 [2290 to 3829] | 2920 [2254 to 3770]

8. Primary Outcome: Chemistry and Hematology Laboratory Measures - Platelets, White Blood Cells (WBC)
Description: For each local laboratory measure, summary statistics are presented by treatment group and timepoint.
Time Frame: Measured at Weeks 0, 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
1000 cells/cubic mm
  WBC (1000 cells/cubic mm)- Week 0: number analyzed (Participants) | 636 | 642 | 642 | 1284
  WBC (1000 cells/cubic mm)- Week 0 | 5.76 [4.8 to 7.1] | 5.76 [4.9 to 6.87] | 6.1 [5.07 to 7.14] | 5.9 [5 to 7.02]
  WBC (1000 cells/cubic mm)- Week 8: number analyzed (Participants) | 618 | 610 | 608 | 1218
  WBC (1000 cells/cubic mm)- Week 8 | 5.72 [4.75 to 6.91] | 5.55 [4.7 to 6.63] | 5.75 [4.92 to 6.99] | 5.63 [4.8 to 6.8]
  WBC (1000 cells/cubic mm)- Week 16: number analyzed (Participants) | 606 | 593 | 586 | 1179
  WBC (1000 cells/cubic mm)- Week 16 | 5.54 [4.57 to 6.9] | 5.53 [4.63 to 6.7] | 5.71 [4.82 to 6.93] | 5.63 [4.72 to 6.83]
  WBC (1000 cells/cubic mm)- Week 24: number analyzed (Participants) | 594 | 586 | 581 | 1167
  WBC (1000 cells/cubic mm)- Week 24 | 5.57 [4.66 to 6.81] | 5.58 [4.66 to 6.64] | 5.6 [4.72 to 6.85] | 5.6 [4.7 to 6.76]
  WBC (1000 cells/cubic mm)- Week 32: number analyzed (Participants) | 576 | 567 | 574 | 1141
  WBC (1000 cells/cubic mm)- Week 32 | 5.6 [4.57 to 6.9] | 5.6 [4.6 to 6.83] | 5.76 [4.84 to 6.91] | 5.69 [4.73 to 6.86]
  WBC (1000 cells/cubic mm)- Week 40: number analyzed (Participants) | 563 | 554 | 556 | 1110
  WBC (1000 cells/cubic mm)- Week 40 | 5.6 [4.65 to 6.71] | 5.6 [4.73 to 6.7] | 5.75 [4.78 to 6.89] | 5.67 [4.77 to 6.81]
  WBC (1000 cells/cubic mm)- Week 48: number analyzed (Participants) | 559 | 543 | 539 | 1082
  WBC (1000 cells/cubic mm)- Week 48 | 5.6 [4.63 to 6.8] | 5.64 [4.77 to 6.7] | 5.79 [4.73 to 7] | 5.69 [4.75 to 6.9]
  WBC (1000 cells/cubic mm)- Week 56: number analyzed (Participants) | 552 | 533 | 538 | 1071
  WBC (1000 cells/cubic mm)- Week 56 | 5.65 [4.67 to 7.01] | 5.54 [4.6 to 6.8] | 5.62 [4.7 to 6.8] | 5.6 [4.67 to 6.8]
  WBC (1000 cells/cubic mm)- Week 64: number analyzed (Participants) | 544 | 529 | 537 | 1066
  WBC (1000 cells/cubic mm)- Week 64 | 5.52 [4.6 to 6.87] | 5.6 [4.65 to 6.54] | 5.62 [4.77 to 6.83] | 5.61 [4.7 to 6.69]
  WBC (1000 cells/cubic mm)- Week 72: number analyzed (Participants) | 540 | 515 | 526 | 1041
  WBC (1000 cells/cubic mm)- Week 72 | 5.57 [4.58 to 6.88] | 5.57 [4.68 to 6.59] | 5.77 [4.73 to 6.89] | 5.66 [4.7 to 6.7]
  Platelets (1000 cells/cubic mm)- Week 0: number analyzed (Participants) | 637 | 640 | 642 | 1282
  Platelets (1000 cells/cubic mm)- Week 0 | 272 [227 to 315] | 275 [234 to 322] | 279 [240 to 323] | 277 [236 to 322]
  Platelets (1000 cells/cubic mm)- Week 8: number analyzed (Participants) | 618 | 609 | 608 | 1217
  Platelets (1000 cells/cubic mm)- Week 8 | 271 [230 to 317] | 275 [234 to 318] | 282 [238 to 323] | 279 [236 to 321]
  Platelets (1000 cells/cubic mm)- Week 16: number analyzed (Participants) | 605 | 591 | 586 | 1177
  Platelets (1000 cells/cubic mm)- Week 16 | 275 [232 to 320] | 275 [235 to 322] | 280 [241 to 329] | 278 [238 to 326]
  Platelets (1000 cells/cubic mm)- Week 24: number analyzed (Participants) | 594 | 585 | 580 | 1165
  Platelets (1000 cells/cubic mm)- Week 24 | 277 [233 to 315] | 278 [233 to 323] | 283 [240 to 330.5] | 280 [238 to 326]
  Platelets (1000 cells/cubic mm)- Week 32: number analyzed (Participants) | 576 | 567 | 574 | 1141
  Platelets (1000 cells/cubic mm)- Week 32 | 272 [231 to 314.5] | 277 [236 to 327] | 285 [243 to 326] | 282 [240 to 327]
  Platelets (1000 cells/cubic mm)- Week 40: number analyzed (Participants) | 564 | 554 | 555 | 1109
  Platelets (1000 cells/cubic mm)- Week 40 | 276 [233 to 324] | 281 [238 to 323] | 285 [241 to 331] | 283 [239 to 329]
  Platelets (1000 cells/cubic mm)- Week 48: number analyzed (Participants) | 559 | 543 | 539 | 1082
  Platelets (1000 cells/cubic mm)- Week 48 | 270 [235 to 320] | 279 [236 to 324] | 282 [246 to 333] | 281 [240 to 329]
  Platelets (1000 cells/cubic mm)- Week 56: number analyzed (Participants) | 552 | 533 | 538 | 1071
  Platelets (1000 cells/cubic mm)- Week 56 | 274 [231 to 324] | 274 [235 to 323] | 280 [238 to 329] | 277 [237 to 326]
  Platelets (1000 cells/cubic mm)- Week 64: number analyzed (Participants) | 544 | 529 | 537 | 1066
  Platelets (1000 cells/cubic mm)- Week 64 | 271.5 [231.5 to 319] | 274 [237 to 325] | 282 [240 to 323] | 277 [238 to 324]
  Platelets (1000 cells/cubic mm)- Week 72: number analyzed (Participants) | 540 | 514 | 526 | 1040
  Platelets (1000 cells/cubic mm)- Week 72 | 274 [234.5 to 326] | 276.5 [238 to 323] | 281 [239 to 329] | 278.5 [238 to 325]

9. Primary Outcome: Chemistry and Hematology Laboratory Measures Meeting Grade 3 AE Criteria or Above
Description: The number (percentage) of participants with chemistry and hematology laboratory measures meeting grade 3 AE criteria or above as specified in the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017] is tabulated by treatment group and timepoint. Excludes measures taken prior to exposure to study product at Week 0/Infusion 1.
Time Frame: Measured at Weeks 8, 16, 24, 32, 40, 48, 56, 64, 72.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
Participants
  ALT (SGPT) (U/L)- Week 8: number analyzed (Participants) | 618 | 612 | 608 | 1220
  ALT (SGPT) (U/L)- Week 8 | 1 | 0 | 2 | 2
  ALT (SGPT) (U/L)- Week 16: number analyzed (Participants) | 606 | 593 | 589 | 1182
  ALT (SGPT) (U/L)- Week 16 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Week 24: number analyzed (Participants) | 594 | 587 | 581 | 1168
  ALT (SGPT) (U/L)- Week 24 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Week 32: number analyzed (Participants) | 577 | 568 | 572 | 1140
  ALT (SGPT) (U/L)- Week 32 | 1 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Week 40: number analyzed (Participants) | 563 | 554 | 554 | 1108
  ALT (SGPT) (U/L)- Week 40 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Week 48: number analyzed (Participants) | 560 | 542 | 539 | 1081
  ALT (SGPT) (U/L)- Week 48 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Week 56: number analyzed (Participants) | 553 | 533 | 538 | 1071
  ALT (SGPT) (U/L)- Week 56 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Week 64: number analyzed (Participants) | 548 | 530 | 536 | 1066
  ALT (SGPT) (U/L)- Week 64 | 1 | 0 | 1 | 1
  ALT (SGPT) (U/L)- Week 72: number analyzed (Participants) | 541 | 514 | 526 | 1040
  ALT (SGPT) (U/L)- Week 72 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 8: number analyzed (Participants) | 618 | 610 | 608 | 1218
  Hemoglobin (g/dL)- Week 8 | 1 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 16: number analyzed (Participants) | 606 | 593 | 586 | 1179
  Hemoglobin (g/dL)- Week 16 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 24: number analyzed (Participants) | 594 | 586 | 581 | 1167
  Hemoglobin (g/dL)- Week 24 | 1 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 32: number analyzed (Participants) | 576 | 567 | 574 | 1141
  Hemoglobin (g/dL)- Week 32 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 40: number analyzed (Participants) | 564 | 554 | 556 | 1110
  Hemoglobin (g/dL)- Week 40 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Week 48: number analyzed (Participants) | 559 | 543 | 539 | 1082
  Hemoglobin (g/dL)- Week 48 | 0 | 1 | 0 | 1
  Hemoglobin (g/dL)- Week 56: number analyzed (Participants) | 553 | 533 | 538 | 1071
  Hemoglobin (g/dL)- Week 56 | 1 | 0 | 1 | 1
  Hemoglobin (g/dL)- Week 64: number analyzed (Participants) | 545 | 529 | 537 | 1066
  Hemoglobin (g/dL)- Week 64 | 0 | 0 | 2 | 2
  Hemoglobin (g/dL)- Week 72: number analyzed (Participants) | 540 | 515 | 526 | 1041
  Hemoglobin (g/dL)- Week 72 | 0 | 0 | 1 | 1
  Creatinine (mg/dL)- Week 8: number analyzed (Participants) | 618 | 612 | 608 | 1220
  Creatinine (mg/dL)- Week 8 | 5 | 1 | 4 | 5
  Creatinine (mg/dL)- Week 16: number analyzed (Participants) | 606 | 593 | 589 | 1182
  Creatinine (mg/dL)- Week 16 | 2 | 3 | 3 | 6
  Creatinine (mg/dL)- Week 24: number analyzed (Participants) | 594 | 587 | 581 | 1168
  Creatinine (mg/dL)- Week 24 | 2 | 4 | 5 | 9
  Creatinine (mg/dL)- Week 32: number analyzed (Participants) | 577 | 568 | 572 | 1140
  Creatinine (mg/dL)- Week 32 | 6 | 2 | 5 | 7
  Creatinine (mg/dL)- Week 40: number analyzed (Participants) | 563 | 554 | 554 | 1108
  Creatinine (mg/dL)- Week 40 | 7 | 2 | 3 | 5
  Creatinine (mg/dL)- Week 48: number analyzed (Participants) | 560 | 542 | 539 | 1081
  Creatinine (mg/dL)- Week 48 | 3 | 0 | 5 | 5
  Creatinine (mg/dL)- Week 56: number analyzed (Participants) | 553 | 533 | 538 | 1071
  Creatinine (mg/dL)- Week 56 | 5 | 2 | 4 | 6
  Creatinine (mg/dL)- Week 64: number analyzed (Participants) | 548 | 530 | 536 | 1066
  Creatinine (mg/dL)- Week 64 | 4 | 1 | 4 | 5
  Creatinine (mg/dL)- Week 72: number analyzed (Participants) | 541 | 514 | 526 | 1040
  Creatinine (mg/dL)- Week 72 | 7 | 1 | 1 | 2
  WBC (1000 cells/cubic mm)- Week 8: number analyzed (Participants) | 618 | 610 | 608 | 1218
  WBC (1000 cells/cubic mm)- Week 8 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)- Week 16: number analyzed (Participants) | 606 | 593 | 586 | 1179
  WBC (1000 cells/cubic mm)- Week 16 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)- Week 24: number analyzed (Participants) | 594 | 586 | 581 | 1167
  WBC (1000 cells/cubic mm)- Week 24 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)- Week 32: number analyzed (Participants) | 576 | 567 | 574 | 1141
  WBC (1000 cells/cubic mm)- Week 32 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)- Week 40: number analyzed (Participants) | 563 | 554 | 556 | 1110
  WBC (1000 cells/cubic mm)- Week 40 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)- Week 48: number analyzed (Participants) | 559 | 543 | 539 | 1082
  WBC (1000 cells/cubic mm)- Week 48 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)- Week 56: number analyzed (Participants) | 552 | 533 | 538 | 1071
  WBC (1000 cells/cubic mm)- Week 56 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)- Week 64: number analyzed (Participants) | 544 | 529 | 537 | 1066
  WBC (1000 cells/cubic mm)- Week 64 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)- Week 72: number analyzed (Participants) | 540 | 515 | 526 | 1041
  WBC (1000 cells/cubic mm)- Week 72 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)- Week 8: number analyzed (Participants) | 618 | 609 | 608 | 1217
  Platelets (1000 cells/cubic mm)- Week 8 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)- Week 16: number analyzed (Participants) | 605 | 591 | 586 | 1177
  Platelets (1000 cells/cubic mm)- Week 16 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)- Week 24: number analyzed (Participants) | 594 | 585 | 580 | 1165
  Platelets (1000 cells/cubic mm)- Week 24 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)- Week 32: number analyzed (Participants) | 576 | 567 | 574 | 1141
  Platelets (1000 cells/cubic mm)- Week 32 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)- Week 40: number analyzed (Participants) | 564 | 554 | 555 | 1109
  Platelets (1000 cells/cubic mm)- Week 40 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)- Week 48: number analyzed (Participants) | 559 | 543 | 539 | 1082
  Platelets (1000 cells/cubic mm)- Week 48 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)- Week 56: number analyzed (Participants) | 552 | 533 | 538 | 1071
  Platelets (1000 cells/cubic mm)- Week 56 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)- Week 64: number analyzed (Participants) | 544 | 529 | 537 | 1066
  Platelets (1000 cells/cubic mm)- Week 64 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)- Week 72: number analyzed (Participants) | 540 | 514 | 526 | 1040
  Platelets (1000 cells/cubic mm)- Week 72 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 8: number analyzed (Participants) | 618 | 610 | 608 | 1218
  Lymphocytes (cells/cubic mm)- Week 8 | 0 | 1 | 0 | 1
  Lymphocytes (cells/cubic mm)- Week 16: number analyzed (Participants) | 606 | 593 | 586 | 1179
  Lymphocytes (cells/cubic mm)- Week 16 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 24: number analyzed (Participants) | 594 | 586 | 581 | 1167
  Lymphocytes (cells/cubic mm)- Week 24 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 32: number analyzed (Participants) | 576 | 567 | 574 | 1141
  Lymphocytes (cells/cubic mm)- Week 32 | 1 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 40: number analyzed (Participants) | 564 | 554 | 556 | 1110
  Lymphocytes (cells/cubic mm)- Week 40 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 48: number analyzed (Participants) | 559 | 543 | 539 | 1082
  Lymphocytes (cells/cubic mm)- Week 48 | 0 | 0 | 1 | 1
  Lymphocytes (cells/cubic mm)- Week 56: number analyzed (Participants) | 552 | 533 | 538 | 1071
  Lymphocytes (cells/cubic mm)- Week 56 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 64: number analyzed (Participants) | 544 | 529 | 537 | 1066
  Lymphocytes (cells/cubic mm)- Week 64 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm)- Week 72: number analyzed (Participants) | 540 | 515 | 526 | 1041
  Lymphocytes (cells/cubic mm)- Week 72 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 8: number analyzed (Participants) | 618 | 610 | 608 | 1218
  Neutrophils (cells/cubic mm)- Week 8 | 0 | 0 | 1 | 1
  Neutrophils (cells/cubic mm)- Week 16: number analyzed (Participants) | 606 | 593 | 586 | 1179
  Neutrophils (cells/cubic mm)- Week 16 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 24: number analyzed (Participants) | 594 | 586 | 581 | 1167
  Neutrophils (cells/cubic mm)- Week 24 | 1 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 32: number analyzed (Participants) | 576 | 567 | 574 | 1141
  Neutrophils (cells/cubic mm)- Week 32 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 40: number analyzed (Participants) | 564 | 554 | 556 | 1110
  Neutrophils (cells/cubic mm)- Week 40 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 48: number analyzed (Participants) | 559 | 543 | 539 | 1082
  Neutrophils (cells/cubic mm)- Week 48 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 56: number analyzed (Participants) | 552 | 533 | 538 | 1071
  Neutrophils (cells/cubic mm)- Week 56 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 64: number analyzed (Participants) | 544 | 529 | 537 | 1066
  Neutrophils (cells/cubic mm)- Week 64 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm)- Week 72: number analyzed (Participants) | 540 | 515 | 526 | 1041
  Neutrophils (cells/cubic mm)- Week 72 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Early Infusion Discontinuation and Reasons for Discontinuation
Description: The number (percentage) of participants with early permanent discontinuation of infusions and their reason for discontinuation is summarized by treatment group. Includes all discontinuations documented on a study case report form.
Time Frame: Measured through Week 72 (the last infusion visit).
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
Participants
  Pregnancy | 2 | 2 | 0 | 2
  HIV infection | 28 | 25 | 15 | 40
  Death | 0 | 0 | 0 | 0
  Clinical event other than reactogenicity | 3 | 16 | 24 | 40
  Reactogenicity Symptom | 0 | 6 | 2 | 8
  Investigator Reason | 4 | 2 | 6 | 8
  Participant refused study product infusion | 2 | 4 | 6 | 10
  Co-enrollment in a study | 1 | 0 | 0 | 0
  Two(2) reactive HIV tests | 1 | 2 | 2 | 4
  Other | 6 | 8 | 10 | 18
  Termination from study for non-medical reason(s) | 30 | 32 | 26 | 58
  No Discontinuation | 560 | 545 | 554 | 1099

11. Primary Outcome: Incidence Rate of Early Infusion Discontinuation
Description: Incidence rate (95% CI) of early infusion discontinuation per 100 person years. Includes discontinuations documented on a study case report form and operational discontinuations defined as 20 consecutive weeks without participant contact. Discontinuations due to pregnancy, death, or HIV-1 infection are right-censored.
Time Frame: Measured through Week 72 (the last infusion visit).
Population: Safety population
Measure: Number (95% Confidence Interval); unit: events per 100 person years
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01
Number analyzed (Participants) | 637 | 642 | 645
events per 100 person years | 5.3 [3.9 to 7.1] | 8.7 [6.9 to 10.9] | 8 [6.3 to 10.2]

12. Primary Outcome: Number of Participants With Documented HIV-1 Infection by the Week 80 Visit
Description: Prevention efficacy (PE) is measured as 1 minus the ratio (VRC01:control) of cumulative incidences of HIV-1 infection diagnosis between enrollment and the week 80 visit for assessment of the primary efficacy end point. Cumulative incidence was estimated with the Nelson-Aalen estimator for the cumulative hazard function, with stratification according to VRC01 dose and trial.
Time Frame: Measured through Week 80.
Population: MITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
Participants | 29 | 28 | 19 | 47
Statistical Analysis 1: Comparison: Placebo vs Pooled VRC01; The primary PE analysis tests the null hypothesis PE equal to zero versus the alternative hypothesis PE not equal to zero using a 2-sided alpha equal 0.05 level Wald test of the equality of log cumulative hazard functions at the week 80 visit for the pooled VRC01 group versus the placebo group; Test type: Other; p = 0.70, wald — The threshold for statistical significance was p = 0.05; Prevention Efficacy (PE) = 8.8, 95% CI 2-sided [-45.1 to 42.6]
Statistical Analysis 2: Comparison: Placebo vs Low-Dose VRC01; A secondary analysis assesses the overall PE of the low-dose VRC01 group versus the placebo group; Test type: Other; Prevention Efficacy (PE) = -9.3, 95% CI 2-sided [-85.3 to 35.5]
Statistical Analysis 3: Comparison: Placebo vs High-Dose VRC01; A secondary analysis assesses the overall PE of the high-dose VRC01 group versus the placebo group; Test type: Other; Prevention Efficacy (PE) = 27.0, 95% CI 2-sided [-30.7 to 59.3]

13. Secondary Outcome: Serum Concentration of VRC01 in Participants Assigned to Receive the mAb
Description: The pharmacokinetic analyses of VRC01 involved a subgroup of VRC01 recipients who had not acquired HIV-1 infection through the week 88 visit and were not likely to have used preexposure prophylaxis (on the basis of self-report or testing of dried blood-spot samples), randomly sampled among the trials and dose groups. Midpoint and trough concentrations are the participant-level median concentrations at the 4-week and 8-week postinfusion visits, respectively, across all 10 infusion intervals.
Time Frame: Day 61 (5 days post infusion #2), Midpoint (4-weeks post infusion visits): Weeks 4, 12, 16, 28, 36, 44, 52, 60, 68, 76 and Trough (infusion visits): Pre dose at Weeks 0 (study entry), 8, 16, 24, 32, 40, 48, 56, 64, and 72.
Population: Pilot study population
Measure: Median (Full Range); unit: μg/ml
Arm/Group | Low-Dose VRC01 | High-Dose VRC01
Number analyzed (Participants) | 12 | 11
μg/ml
  4-week post infusion visit | 19.8 [12.7 to 27.2] | 44.7 [29.4 to 80.5]
  8-week post infusion visit | 4.7 [1.5 to 6] | 8.3 [2.3 to 16.7]
  Day 61 | 88.9 [38.3 to 111.1] | 257.9 [158.6 to 327.5]

14. Secondary Outcome: VRC01 Clinical Lot Neutralization of Founder Viruses (IC80)
Description: The VRC01 80% inhibitory concentration (IC80) of acquired isolates was measured with the TZM-bl assay using the earliest available post-HIV-infection serum sample. Median and IQR are summarized immediately below, then the analysis of prevention efficacy was repeated for each of three prespecified categories of in vitro susceptibility of the infecting strain (IC80 less than 1 μg per milliliter, 1 to 3 μg per milliliter, or >3 μg per milliliter) with the use of the Aalen-Johansen estimator.
Time Frame: Measured through Week 80.
Population: MITT population
Measure: Median (Inter-Quartile Range); unit: μg/ml
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
Number analyzed (Participants) | 637 | 642 | 645 | 1287
μg/ml | 4.39 [1.37 to 30.74] | 4.54 [2.7 to 100] | 22.8 [3.64 to 100] | 5.32 [2.96 to 100]
Statistical Analysis 1: Comparison: Placebo vs Pooled VRC01; PE against IC80 of least sensitive variant less than 1; Test type: Other; Prevention Efficacy (PE) = 78.6, 95% CI 2-sided [17.3 to 94.4]
Statistical Analysis 2: Comparison: Placebo vs Pooled VRC01; PE against IC80 of least sensitive variant 1-3; Test type: Other; Prevention Efficacy (PE) = 7.4, 95% CI 2-sided [-187.5 to 70.2]
Statistical Analysis 3: Comparison: Placebo vs Pooled VRC01; PE against IC80 of least sensitive variant > 3; Test type: Other; Prevention Efficacy (PE) = -1.9, 95% CI 2-sided [-83.1 to 43.3]

15. Secondary Outcome: VRC01 Serum Neutralization of Autologous Founder Viruses (ID50, ID80)
Description: Autologous titer (ID50, ID80) summaries, based on most sensitive virus, for first RNA+ samples from a subset of HIV-infected VRC01 recipients. Values below the limit of detection (less than 10) were set to NA. Summaries are only computed for the Pooled VRC01 arm.
Time Frame: First RNA+ Sample detected from baseline up to Week 104.
Population: Subset of HIV-infected VRC01 recipients
Measure: Median (Full Range); unit: titer
Arm/Group | Pooled VRC01
Number analyzed (Participants) | 23
titer
  ID50 | NA [NA to 34.51] — Values below the limit of detection (less than 10) were set to NA.
  ID80 | NA [NA to 12.77] — Values below the limit of detection (less than 10) were set to NA.

ADVERSE EVENTS:
Time Frame: The AE reporting period for this study comprises the entire study period for each individual participant (from study enrollment until study completion at the week 104 visit or discontinuation of the study)
Arm/Group | Placebo | Low-Dose VRC01 | High-Dose VRC01 | Pooled VRC01
All-Cause Mortality (participants affected / at risk) | 1/637 | 2/642 | 0/645 | 2/1287
Serious Adverse Events (participants affected / at risk) | 26/637 | 10/642 | 23/645 | 33/1287
Other Adverse Events (participants affected / at risk) | 594/637 | 587/642 | 591/645 | 1178/1287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=637) | Low-Dose VRC01 (N=642) | High-Dose VRC01 (N=645) | Pooled VRC01 (N=1287)
Any Event in SOC (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Infections and infestations) | 5 (5) | 4 (4) | 8 (8) | 12 (12)
Abortion infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis gonococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malaria (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 6 (6) | 8 (8)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Uterine injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Pregnancy, puerperium and perinatal conditions) | 7 (8) | 3 (3) | 5 (5) | 8 (8)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
False labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=637) | Low-Dose VRC01 (N=642) | High-Dose VRC01 (N=645) | Pooled VRC01 (N=1287)
Any Event in SOC (Blood and lymphatic system disorders) | 12 (15) | 15 (21) | 17 (21) | 32 (42)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 2 (2) | 3 (3) | 5 (5)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 4 (4) | 6 (6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (6) | 3 (4) | 7 (10)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 4 (5) | 6 (7)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Normochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0) | 2 (3)
Any Event in SOC (Cardiac disorders) | 2 (2) | 3 (3) | 5 (5) | 8 (8)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 3 (3) | 3 (3) | 6 (6)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Ear and labyrinth disorders) | 10 (11) | 8 (8) | 9 (9) | 17 (17)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 5 (6) | 5 (5) | 5 (5) | 10 (10)
External ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Any Event in SOC (Eye disorders) | 42 (52) | 25 (28) | 25 (28) | 50 (56)
Asthenopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Astigmatism (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 19 (23) | 16 (18) | 11 (12) | 27 (30)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 5 (6) | 3 (3) | 3 (3) | 6 (6)
Eye pruritus (Eye disorders) | 2 (2) | 3 (3) | 5 (5) | 8 (8)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelids pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gaze palsy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermetropia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periorbital pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presbyopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pterygium (Eye disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Refraction disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Gastrointestinal disorders) | 220 (325) | 161 (273) | 190 (309) | 351 (582)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 49 (55) | 26 (31) | 30 (33) | 56 (64)
Abdominal pain lower (Gastrointestinal disorders) | 32 (35) | 17 (19) | 27 (30) | 44 (49)
Abdominal pain upper (Gastrointestinal disorders) | 9 (9) | 7 (10) | 7 (7) | 14 (17)
Anal fissure (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 3 (3)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 2 (6) | 0 (0) | 2 (6)
Constipation (Gastrointestinal disorders) | 18 (18) | 11 (12) | 18 (20) | 29 (32)
Dental caries (Gastrointestinal disorders) | 7 (7) | 11 (11) | 9 (11) | 20 (22)
Diarrhoea (Gastrointestinal disorders) | 34 (42) | 27 (29) | 37 (48) | 64 (77)
Duodenogastric reflux (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 26 (31) | 34 (42) | 30 (34) | 64 (76)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 24 (26) | 22 (26) | 29 (35) | 51 (61)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 (12) | 13 (14) | 14 (15) | 27 (29)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 7 (8) | 2 (2) | 3 (3) | 5 (5)
Hyperaesthesia teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 2 (2) | 6 (8) | 3 (5) | 9 (13)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 6 (6) | 3 (3) | 9 (9)
Nausea (Gastrointestinal disorders) | 19 (21) | 13 (13) | 15 (18) | 28 (31)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue geographic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 20 (21) | 20 (22) | 20 (22) | 40 (44)
Trichoglossia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 12 (12) | 6 (6) | 8 (8) | 14 (14)
Any Event in SOC (General disorders) | 131 (186) | 137 (211) | 131 (185) | 268 (396)
Adverse drug reaction (General disorders) | 3 (3) | 2 (2) | 5 (6) | 7 (8)
Asthenia (General disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Chest pain (General disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (3) | 5 (5) | 7 (8)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hangover (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 100 (142) | 112 (176) | 94 (134) | 206 (310)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Infusion site pruritus (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Malaise (General disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Mass (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nodule (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 9 (9) | 10 (11) | 10 (11) | 20 (22)
Oedema peripheral (General disorders) | 2 (3) | 0 (0) | 2 (2) | 2 (2)
Pain (General disorders) | 4 (5) | 5 (5) | 7 (7) | 12 (12)
Peripheral swelling (General disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 5 (5) | 7 (7)
Suprapubic pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Hepatobiliary disorders) | 2 (2) | 1 (5) | 1 (1) | 2 (6)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatty liver alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (5) | 0 (0) | 1 (5)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Immune system disorders) | 3 (3) | 10 (10) | 7 (8) | 17 (18)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Atopy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Food allergy (Immune system disorders) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 3 (3) | 3 (3) | 6 (6)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Infections and infestations) | 474 (1458) | 481 (1535) | 487 (1560) | 968 (3095)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 4 (4)
Abscess limb (Infections and infestations) | 11 (12) | 9 (9) | 5 (6) | 14 (15)
Abscess of eyelid (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 9 (12) | 19 (24) | 14 (16) | 33 (40)
Acute sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Alveolar osteitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Bacterial diarrhoea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial food poisoning (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 22 (23) | 15 (17) | 20 (20) | 35 (37)
Bartholin's abscess (Infections and infestations) | 0 (0) | 2 (3) | 2 (2) | 4 (5)
Blister infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 32 (41) | 24 (27) | 19 (24) | 43 (51)
Breast abscess (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 14 (15) | 7 (9) | 7 (9) | 14 (18)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bullous impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Burn infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 2 (2) | 1 (2) | 3 (4)
Cellulitis (Infections and infestations) | 8 (9) | 5 (5) | 4 (5) | 9 (10)
Cervicitis (Infections and infestations) | 1 (2) | 1 (1) | 4 (4) | 5 (5)
Chlamydial infection (Infections and infestations) | 7 (7) | 6 (6) | 6 (6) | 12 (12)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 14 (17) | 21 (25) | 14 (17) | 35 (42)
Conjunctivitis bacterial (Infections and infestations) | 5 (5) | 0 (0) | 2 (2) | 2 (2)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cutaneous larva migrans (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Cystitis escherichia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dermatophytosis (Infections and infestations) | 9 (11) | 14 (21) | 5 (7) | 19 (28)
Dermatophytosis of nail (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 2 (3)
Diarrhoea infectious (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Dysentery (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ear infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Eye abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (4) | 3 (5)
Folliculitis (Infections and infestations) | 11 (11) | 18 (19) | 14 (16) | 32 (35)
Fungal infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Fungal skin infection (Infections and infestations) | 17 (18) | 14 (15) | 6 (9) | 20 (24)
Furuncle (Infections and infestations) | 5 (8) | 6 (7) | 11 (16) | 17 (23)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 58 (69) | 61 (72) | 52 (67) | 113 (139)
Gastroenteritis bacterial (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Genital abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Genital candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Genital herpes (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 5 (5)
Genital herpes simplex (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Genital ulcer syndrome (Infections and infestations) | 4 (4) | 10 (10) | 4 (4) | 14 (14)
Genitourinary chlamydia infection (Infections and infestations) | 131 (166) | 144 (172) | 148 (193) | 292 (365)
Genitourinary tract gonococcal infection (Infections and infestations) | 50 (54) | 59 (70) | 54 (65) | 113 (135)
Genitourinary tract infection (Infections and infestations) | 2 (2) | 4 (4) | 2 (2) | 6 (6)
Gingivitis (Infections and infestations) | 5 (5) | 2 (2) | 2 (2) | 4 (4)
Gonococcal infection (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 5 (5)
Gonorrhoea (Infections and infestations) | 2 (2) | 1 (1) | 4 (4) | 5 (5)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helminthic infection (Infections and infestations) | 4 (4) | 4 (4) | 2 (2) | 6 (6)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 2 (2) | 1 (1) | 4 (4) | 5 (5)
Impetigo (Infections and infestations) | 5 (5) | 4 (5) | 4 (4) | 8 (9)
Infected skin ulcer (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 6 (7) | 5 (5) | 6 (7) | 11 (12)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Laryngitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 17 (17) | 16 (17) | 11 (14) | 27 (31)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 23 (33) | 15 (20) | 17 (22) | 32 (42)
Mastitis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 4 (4)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Mumps (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 20 (22) | 18 (20) | 17 (20) | 35 (40)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Oral herpes (Infections and infestations) | 12 (17) | 5 (5) | 8 (8) | 13 (13)
Oral viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 4 (4) | 4 (4) | 5 (6) | 9 (10)
Otitis media (Infections and infestations) | 8 (11) | 10 (11) | 9 (10) | 19 (21)
Otitis media acute (Infections and infestations) | 0 (0) | 3 (3) | 2 (4) | 5 (7)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 15 (17) | 10 (12) | 12 (14) | 22 (26)
Perineal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 27 (29) | 22 (26) | 36 (43) | 58 (69)
Pharyngitis bacterial (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 6 (6)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Rash pustular (Infections and infestations) | 1 (1) | 2 (2) | 1 (2) | 3 (4)
Respiratory tract infection (Infections and infestations) | 12 (13) | 12 (12) | 9 (9) | 21 (21)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 4 (4) | 6 (6) | 10 (10)
Rhinitis (Infections and infestations) | 12 (15) | 11 (14) | 10 (13) | 21 (27)
Salmonellosis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Schistosomiasis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Secondary syphilis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sexually transmitted disease (Infections and infestations) | 3 (3) | 2 (2) | 5 (6) | 7 (8)
Sinusitis (Infections and infestations) | 9 (9) | 11 (16) | 6 (6) | 17 (22)
Skin bacterial infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 13 (13) | 15 (18) | 16 (19) | 31 (37)
Syphilis (Infections and infestations) | 10 (10) | 13 (13) | 12 (13) | 25 (26)
Syphilis genital (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Systemic bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinea capitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Tinea faciei (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Tinea infection (Infections and infestations) | 10 (11) | 4 (5) | 5 (5) | 9 (10)
Tinea manuum (Infections and infestations) | 3 (4) | 1 (1) | 1 (2) | 2 (3)
Tinea pedis (Infections and infestations) | 2 (2) | 2 (2) | 1 (2) | 3 (4)
Tinea versicolour (Infections and infestations) | 13 (15) | 9 (12) | 10 (10) | 19 (22)
Tonsillitis (Infections and infestations) | 31 (37) | 39 (45) | 50 (65) | 89 (110)
Tonsillitis bacterial (Infections and infestations) | 2 (2) | 9 (11) | 3 (3) | 12 (14)
Tooth abscess (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 6 (6)
Trichomoniasis (Infections and infestations) | 6 (7) | 5 (5) | 6 (7) | 11 (12)
Typhoid fever (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 160 (276) | 186 (315) | 169 (300) | 355 (615)
Upper respiratory tract infection bacterial (Infections and infestations) | 5 (5) | 6 (8) | 5 (8) | 11 (16)
Urethritis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Urethritis chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urethritis gonococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 87 (116) | 88 (119) | 96 (131) | 184 (250)
Urinary tract infection bacterial (Infections and infestations) | 10 (12) | 10 (12) | 9 (9) | 19 (21)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urogenital infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urogenital trichomoniasis (Infections and infestations) | 8 (12) | 20 (25) | 24 (27) | 44 (52)
Vaginal infection (Infections and infestations) | 5 (5) | 9 (9) | 5 (5) | 14 (14)
Vaginitis chlamydial (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Varicella (Infections and infestations) | 4 (4) | 5 (5) | 1 (1) | 6 (6)
Viral infection (Infections and infestations) | 1 (1) | 2 (2) | 4 (4) | 6 (6)
Viral rhinitis (Infections and infestations) | 8 (9) | 0 (0) | 4 (5) | 4 (5)
Viral upper respiratory tract infection (Infections and infestations) | 13 (16) | 15 (18) | 16 (21) | 31 (39)
Vulval abscess (Infections and infestations) | 2 (3) | 1 (1) | 5 (6) | 6 (7)
Vulvovaginal candidiasis (Infections and infestations) | 51 (67) | 45 (55) | 52 (57) | 97 (112)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Vulvovaginitis (Infections and infestations) | 8 (14) | 7 (10) | 9 (10) | 16 (20)
Vulvovaginitis gonococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginitis trichomonal (Infections and infestations) | 36 (42) | 38 (54) | 50 (68) | 88 (122)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound sepsis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Any Event in SOC (Injury, poisoning and procedural complications) | 91 (103) | 99 (136) | 85 (101) | 184 (237)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 6 (6) | 14 (19) | 6 (6) | 20 (25)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 7 (8) | 3 (3) | 10 (11)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Eye injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Face injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 6 (6) | 8 (8)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Foreign body in reproductive tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 2 (2) | 6 (6) | 2 (3) | 8 (9)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Induced abortion haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 9 (10) | 22 (28) | 15 (17) | 37 (45)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 6 (6) | 3 (3) | 1 (1) | 4 (4)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 6 (8) | 3 (3) | 9 (11)
Limb injury (Injury, poisoning and procedural complications) | 6 (6) | 5 (5) | 7 (7) | 12 (12)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 9 (9) | 5 (5) | 7 (7) | 12 (12)
Skin abrasion (Injury, poisoning and procedural complications) | 6 (6) | 3 (3) | 4 (4) | 7 (7)
Skin laceration (Injury, poisoning and procedural complications) | 6 (6) | 6 (6) | 4 (4) | 10 (10)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 8 (8) | 8 (8) | 9 (12) | 17 (20)
Splinter (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 9 (9) | 6 (6) | 3 (3) | 9 (9)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Investigations) | 236 (436) | 220 (372) | 227 (406) | 447 (778)
Alanine aminotransferase increased (Investigations) | 60 (88) | 39 (48) | 59 (81) | 98 (129)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 8 (11) | 2 (2) | 3 (6) | 5 (8)
Bilirubin conjugated increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Bilirubin urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Blood creatine increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Blood creatinine increased (Investigations) | 88 (133) | 91 (121) | 96 (126) | 187 (247)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 2 (3)
Blood pressure decreased (Investigations) | 3 (4) | 8 (8) | 5 (5) | 13 (13)
Blood pressure increased (Investigations) | 40 (59) | 47 (75) | 43 (64) | 90 (139)
Body temperature decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Carbon dioxide decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac murmur (Investigations) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Fungal test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 42 (62) | 43 (66) | 39 (69) | 82 (135)
Heart rate increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 1 (2)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 3 (3) | 3 (3) | 6 (6)
Neutrophil count decreased (Investigations) | 22 (32) | 9 (10) | 13 (14) | 22 (24)
Platelet count decreased (Investigations) | 15 (19) | 10 (13) | 10 (16) | 20 (29)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Red blood cells urine (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Smear vaginal abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 5 (5) | 4 (4) | 9 (9)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 4 (5) | 2 (3) | 4 (4) | 6 (7)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Metabolism and nutrition disorders) | 33 (42) | 34 (46) | 46 (54) | 80 (100)
Abnormal loss of weight (Metabolism and nutrition disorders) | 5 (7) | 10 (14) | 12 (15) | 22 (29)
Decreased appetite (Metabolism and nutrition disorders) | 19 (22) | 20 (25) | 22 (26) | 42 (51)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperphagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2) | 3 (4)
Iron deficiency (Metabolism and nutrition disorders) | 7 (7) | 2 (2) | 9 (9) | 11 (11)
Polydipsia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 135 (191) | 117 (170) | 132 (186) | 249 (356)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (33) | 23 (27) | 23 (26) | 46 (53)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 61 (75) | 51 (64) | 55 (73) | 106 (137)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 5 (5)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 0 (0) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (9) | 4 (4) | 3 (3) | 7 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 13 (15) | 12 (12) | 25 (27)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (17) | 11 (13) | 16 (17) | 27 (30)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 10 (10) | 15 (15) | 25 (25)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (9) | 6 (6) | 14 (15)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (13) | 12 (13) | 21 (22) | 33 (35)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 4 (4) | 7 (7) | 11 (11)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2) | 2 (2) | 4 (4)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Any Event in SOC (Nervous system disorders) | 156 (223) | 145 (206) | 143 (220) | 288 (426)
Dizziness (Nervous system disorders) | 26 (26) | 18 (22) | 17 (19) | 35 (41)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 121 (167) | 123 (162) | 118 (182) | 241 (344)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Hyposmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Meningism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 6 (6) | 0 (0) | 4 (4) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Syncope (Nervous system disorders) | 4 (5) | 2 (3) | 2 (2) | 4 (5)
Tension headache (Nervous system disorders) | 5 (5) | 6 (7) | 9 (9) | 15 (16)
Tremor (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Ulnar nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Pregnancy, puerperium and perinatal conditions) | 6 (8) | 10 (11) | 13 (14) | 23 (25)
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 8 (9) | 11 (11) | 19 (20)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Psychiatric disorders) | 17 (20) | 18 (21) | 20 (23) | 38 (44)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3) | 5 (5) | 8 (8)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 5 (6) | 3 (3) | 8 (9)
Emotional distress (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (5) | 4 (4) | 6 (7) | 10 (11)
Libido decreased (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Loss of libido (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pica (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Psychogenic pseudosyncope (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 2 (2) | 2 (2) | 3 (3) | 5 (5)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Terminal insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Renal and urinary disorders) | 63 (86) | 80 (100) | 60 (75) | 140 (175)
Crystalluria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cystitis interstitial (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 14 (15) | 10 (10) | 8 (9) | 18 (19)
Glycosuria (Renal and urinary disorders) | 3 (3) | 1 (1) | 3 (4) | 4 (5)
Haematuria (Renal and urinary disorders) | 12 (14) | 28 (28) | 12 (13) | 40 (41)
Ketonuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Polyuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Proteinuria (Renal and urinary disorders) | 42 (49) | 52 (56) | 37 (42) | 89 (98)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Reproductive system and breast disorders) | 174 (262) | 174 (246) | 142 (205) | 316 (451)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 48 (63) | 44 (65) | 48 (58) | 92 (123)
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adnexa uteri pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Breast discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Breast mass (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 3 (3) | 4 (4)
Breast pain (Reproductive system and breast disorders) | 7 (7) | 8 (9) | 5 (6) | 13 (15)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Coital bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 15 (18) | 15 (16) | 7 (7) | 22 (23)
Dyspareunia (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 3 (3) | 4 (4)
Galactorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Genital blister (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Genital pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Genital ulceration (Reproductive system and breast disorders) | 3 (3) | 3 (3) | 3 (3) | 6 (6)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 2 (2) | 4 (4) | 4 (5) | 8 (9)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Menometrorrhagia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nipple inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 9 (10) | 5 (5) | 5 (5) | 10 (10)
Perineal rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polymenorrhoea (Reproductive system and breast disorders) | 1 (1) | 2 (3) | 1 (1) | 3 (4)
Uterine cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Vaginal discharge (Reproductive system and breast disorders) | 97 (126) | 90 (114) | 70 (87) | 160 (201)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Vaginal ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulval ulceration (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 10 (11) | 6 (6) | 7 (7) | 13 (13)
Vulvovaginal rash (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vulvovaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Withdrawal bleed (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 71 (83) | 57 (62) | 49 (58) | 106 (120)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (2) | 3 (4)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (45) | 21 (21) | 22 (26) | 43 (47)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (3) | 7 (7)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 6 (6) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 11 (11) | 7 (7) | 18 (18)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 10 (11) | 5 (5) | 15 (16)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 121 (154) | 143 (190) | 125 (173) | 268 (363)
Acne (Skin and subcutaneous tissue disorders) | 11 (12) | 6 (6) | 11 (12) | 17 (18)
Acne cystic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 11 (13) | 6 (9) | 5 (6) | 11 (15)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 7 (7) | 8 (9) | 8 (8) | 16 (17)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 1 (1) | 5 (5)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6) | 12 (13) | 18 (19)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 9 (10) | 13 (18) | 10 (15) | 23 (33)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Keloid scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Miliaria (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) | 3 (3) | 6 (7)
Papule (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 3 (3) | 5 (5)
Pityriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (27) | 33 (36) | 23 (27) | 56 (63)
Rash (Skin and subcutaneous tissue disorders) | 22 (25) | 19 (24) | 16 (19) | 35 (43)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (3) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4) | 2 (2) | 6 (6)
Rash papular (Skin and subcutaneous tissue disorders) | 14 (14) | 14 (15) | 16 (18) | 30 (33)
Rash pruritic (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (9) | 8 (8) | 15 (17)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 16 (16) | 19 (19) | 35 (35)
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Social circumstances) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Victim of sexual abuse (Social circumstances) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Any Event in SOC (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Finger amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Vascular disorders) | 5 (6) | 12 (17) | 13 (16) | 25 (33)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 4 (5) | 10 (15) | 10 (12) | 20 (27)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vascular pain (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT02568215/Prot_001.pdf
  • Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT02568215/SAP_002.pdf
  • Informed Consent Form (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT02568215/ICF_000.pdf